CLINICAL TRIAL: NCT06222177
Title: Defining High-resolution Manometry Thresholds of Backward Pressure Across the Lower Esophageal Sphincter Through Straight Leg Raise Maneuver in Obese Patients
Brief Title: Thresholds of SLR Maneuver in Obese Patients
Acronym: SLR obese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Medical University of Vienna (Other); University of Campania Luigi Vanvitelli (Other); Università Vita-Salute San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: SLR_Obese
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GERD group: Patients with AET>6% at pH-study
  Interventions: Diagnostic Test: Pathophysiologic evaluation
- Non GERD group: Patients with AET<6% at pH-study
  Interventions: Diagnostic Test: Pathophysiologic evaluation

INTERVENTIONS:
Diagnostic Test: Pathophysiologic evaluation — High-resolution manometry and pH study

SUMMARY:
There is an increasing interest in High resolution manometry (HRM) in the preoperative assessment of patients with obesity, in order to identify the best surgical option. Sleeve gastrectomy (SG) has been known to increase the risk of gastro-esophageal reflux disease (GERD). Different techniques have been recently developed and validated to offer to these patients protection against pathologic GERD after SG.

A recent study found a significant correlation between straight leg raise (SLR) maneuver during HRM and a positive pH-study. However, these maneuver has not been validated in an obese population, therefore the normality cut-off remain unknown.

A multicenter study with a large number of patients undergoing pre-operative assessment for bariatric surgery could provide a precise threshold to predict pathologic esophageal acid exposure time.

ELIGIBILITY:
Inclusion Criteria:

* Complete and adequate HRM and pH-impedance study performed within 2 weeks
* Successfully performed SLR maneuver (adequate intra-abdominal pressure augmentation)
* Obese with BMI>35 Kg/m2

Exclusion Criteria:

* Patients under the age of 18
* Patients with prior foregut surgery
* Paraesophageal hiatal hernia
* Scleroderma
* Eosinophilic esophagitis
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with thorough pathophysiologic evaluation with or without suspect of GERD
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Acid exposure time | January-March 2024

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonaldi M, Rubicondo C, Andreasi V, Giorgi R, Cesana G, Ciccarese F, Uccelli M, Zanoni A, Villa R, De Carli S, Oldani A, Dokic D, Olmi S. Role of Preoperative High-Resolution Manometry in the Identification of Patients at High Risk of Postoperative GERD Symptoms 1 Year After Sleeve Gastrectomy. Obes Surg. 2023 Sep;33(9):2749-2757. doi: 10.1007/s11695-023-06732-x. Epub 2023 Jul 19. PMID 37466827
- [Result] Memon MA, Osland E, Yunus RM, Alam K, Hoque Z, Khan S. Gastroesophageal reflux disease following laparoscopic vertical sleeve gastrectomy and laparoscopic roux-en-Y gastric bypass: meta-analysis and systematic review of 5-year data. Dis Esophagus. 2024 Feb 29;37(3):doad063. doi: 10.1093/dote/doad063. PMID 37935430
- [Result] Siboni S, Kristo I, Rogers BD, De Bortoli N, Hobson A, Louie B, Lee YY, Tee V, Tolone S, Marabotto E, Visaggi P, Haworth J, Ivy M, Greenan G, Facchini C, Masuda T, Yano F, Perry K, Balasubramanian G, Theodorou D, Triantafyllou T, Cusmai L, Boveri S, Schoppmann SF, Gyawali CP, Bonavina L. Improving the Diagnostic Yield of High-Resolution Esophageal Manometry for GERD: The "Straight Leg-Raise" International Study. Clin Gastroenterol Hepatol. 2023 Jul;21(7):1761-1770.e1. doi: 10.1016/j.cgh.2022.10.008. Epub 2022 Oct 19. PMID 36270615